CLINICAL TRIAL: NCT07211217
Title: Time Restricted Eating (TRE) in Bipolar Disorder
Acronym: TREBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Associate Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P002114
Record Dates: First submitted 2025-09-26; First posted 2025-10-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder (BD); Bipolar Disorder Depression; Overweight (BMI > 30)
Keywords: Time Restricted Eating
MeSH Terms: conditions — Bipolar Disorder; Overweight; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Waitlist Control Group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restrictive Eating Condition (Active Comparator): TRE is a dietary intervention where participants eat all of their food within a specific 8-hour eating window, for example eating only between 10am and 6pm. Participants will not be asked to change what they eat, only when to eat. Participants will keep a daily Food Timing Log to record the time of the first and last food and drink that they consume each day. The study will ask participants to continue to do this daily throughout the study (~8 weeks).
  Interventions: Other: Time Restricted Eating
- Waitlist Condition (No Intervention): Participants assigned to the wait list condition will have the option of receiving the TRE intervention after 20 weeks.

INTERVENTIONS:
Other: Time Restricted Eating — See arms description
  Arms: Time Restrictive Eating Condition

SUMMARY:
This is a randomized controlled trial investigating the effects of an 8-TRE intervention compared to a wait list (control) on metabolic health and body composition in people diagnosed with BD and who are currently obese and at least mildly depressed. Following a 1-week baseline assessment, participants will be randomized to either a TRE or the wait list (1-to-1 ratio) for 8 weeks. At baseline, Week 8 (post treatment), and Week 20 (follow-up), investigators will assess daily eating patterns for one week, followed by collection of fasting lipids, body weight and vital signs. At Week 4 (i.e., mid-treatment), the investigators will assess self-reported outcomes only. Participants assigned to the wait list condition will have the option of receiving the TRE intervention after 20 weeks.

DETAILED DESCRIPTION:
The overall goal of this study is to examine the effects of TRE on weight loss and secondary health outcomes in individuals with BD,. A secondary goal is to determine whether these effects are mediated by improvements in circadian rhythms.

Using an 8-week trial of 8-hour TRE compared to a wait list control group, the study will test the following specific aims:

* Examine the effect TRE on weight loss
* if compared to wait list control, individuals assigned to TRE will have greater improvement in waist circumference, depression, anxiety, cognition, sleep and daily functioning.
* if a change in circadian timing will significantly mediate the degree of improvement in body weight with TRE.

Our sample will be representative of the target population, or adults with bipolar disorder who are currently obese and depressed. The study interventions will be offered via telehealth to reduce barriers to access (e.g., childcare, time, parking/transportation costs, less time out of work).

Participants will have a study visit at the start (week 0), midway through (week 4), at the end of the 8-week intervention (week 8), and at a 3-month follow-up (week 20). Study visits will occur after 7 days of monitoring their food intake on Meallogger. To accommodate for scheduling conflicts that may arise, these visits can occur within +3 days of their scheduled dates, if necessary. Study procedures conducted during and surrounding these visits are the same for Weeks 0, 8 and 20.

To recognize participants for the time and effort involved in completing all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18-65 years)
* Diagnosed with bipolar disorder (i.e., subtype Bipolar I or II as assessed with the Quick SCID)21
* Currently experiencing depression (i.e., PHQ-9 ≥ 10)22
* Currently overweight (i.e., Body mass index (BMI) > 30 kg/m2)
* Provides Informed Consent

Exclusion Criteria:

1. Dietary factors:

   1. Diagnosis, or strong clinical suspicion, of eating disorders, including but not limited to, anorexia nervosa, bulimia nervosa, binge eating disorder (as assessed with the Quick SCID)
   2. Concurrent dietary intervention or modification unrelated to study procedures
2. Psychiatric factors:

   1. Severe depression (i.e., PHQ-9>20)
   2. Experiencing manic symptoms (i.e., ASRM < 6)23
   3. Active suicidal ideation (i.e., PHQ-9, item 9 >2)
   4. Current alcohol/substance use disorder (as assessed with the Quick SCID)
3. Medical factors:

   1. Use of weight loss medications or supplements
   2. Use of medications that may cause weight loss or gain, unless body weight and medication usage remained stable for at least 6 months
   3. Previous weight loss surgery
   4. Malignancy within past 2 years
   5. Major surgery within past 3 months
   6. Medical instability considered to interfere with study procedures
   7. Use of medications that have the potential to cause hypoglycemia (e.g., insulin, sulfonylureas)
   8. Undergoing treatment for cancer
   9. Use of medications for which time restricted eating would interfere with recommended timing of medication ingestion with food intake.
4. Lifestyle and other factors:

   a. Work or social schedules that would impede ability to adhere to study protocol
5. Adherence factors:

   1. Ability to adhere to study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | Week 0, Week 8, Week 20
  Body weight will be collected in the fasted state using a digital scale (lbs)

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Week 0, Week 4, Week 8, Week 20
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Generalized Anxiety Disorder scale (GAD-7) | Week 0, Week 4, Week 8 and Week 20
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item questionnaire that is used to measure or assess the severity of generalized anxiety disorder (GAD). The GAD-7 has good reliability, criterion, construct, factorial, and procedural validity. The raw score ranges from 0 to 21. Increasing scores are associated with multiple domains of functional impairment. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Pittsburgh Sleep Quality Index (PSQI) | Week 0, Week 4, Week 8, Week 20
  Change in sleep quality as measure by the Pittsburgh Sleep Quality Index (PSQI) global score. PSQI global score range is 0-21 with higher scores indicating more sleep disturbance. The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A global PSQI score greater than 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% in distinguishing good and poor sleepers.
Cognitive complaints in bipolar disorder rating assessment (COBRA) | Week 0, Week 4, Week 8, Week 20
  The Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) evaluates cognitive impairments which were perceived in daily living. It consists of 16-items using a 4-point Likert scale as follows for each item: 0 = never, 1 = sometimes, 2 = often, and 3 = always. The COBRA had a one-factor structure and showed high internal consistency.
Patient-reported Outcome Measurement Information System (PROMIS) Cognitive Function Short Form 8a | Week 0, Week 4, Week 8, Week 20
  Patient-reported Outcome Measurement Information System (PROMIS) Cognitive Function Short Form 8a is an 8-item self report questionnaire assess subjective cognitive difficulties regarding a patient's concentration, memory, language, mental acuity, as well as perceived changes in cognitive functioning. It has strong internal consistency reliability, supporting its use as a reliable measure of subjective cognitive functioning. This measure has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance). The scale includes four items per domain, each scored from 1 to 5. The scale also includes one question at the end about pain intensity, which is scored from 0 to 10. The possible score ranges from 8 to 40. Higher scores indicate poorer outcomes.
World Health Organization Disability Assessment Scale (WHODAS 2.0) | Week 0, Week 4, Week 8, Week 20
  The adult self-administered version of the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 36-item measure that assesses disability in adults age 18 years and older. It assesses disability across six domains, including understanding and communicating, getting around, self-care, getting along with people, life activities (i.e., household, work, and/or school activities), and participation in society. Each item is rated on a 5-point scale from 0 (none) to 4 (extreme or cannot do), with higher scores indicating greater disability. The total score is calculated by summing the item scores, which can then be converted into a standardized score ranging from 0 to 100, with higher scores indicating greater disability.
The Altman Self-Rating Mania Scale (ASRM) | Week 0, Week 4, Week 8, Week 20
  The Altman Self-Rating Mania Scale (ASRM) is a five-item scale that assesses mood, self-confidence, sleep disturbance, speech, and activity level over a week. The ASRM at a screening cutoff score of 5.5 has shown an optimal combination of sensitivity and specificity (85% and 86%, respectively). The ASRM score range from 5 to 25 with higher scores indicating greater severity of manic symptoms
Changes in waist size | Week 0, 8, and 20
  Measurements of the waist

CONTACTS AND LOCATIONS:
Overall Officials: Louisa G. Sylvia, PhD, Principal Investigator — Massachusetts General Hospital